CLINICAL TRIAL: NCT00651157
Title: A Phase II Trial of Intravenous Administration of Reovirus Serotype 3 - Dearing Strain (Reolysin®) in Patients With Metastatic Melanoma
Brief Title: Viral Therapy in Treating Patients With Metastatic Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00233; NCI-2009-00233 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MAYO-MC0672; 7848; CDR0000592801; MC0672 (Other: Mayo Clinic); 7848 (Other: CTEP); N01CM00070 (NIH)
Record Dates: First submitted 2008-04-01; First posted 2008-04-02 (Estimated); Results first posted 2013-10-16 (Estimated); Last update posted 2014-04-22 (Estimated); Status verified 2014-02

CONDITIONS: Recurrent Melanoma; Stage IV Melanoma
MeSH Terms: conditions — Melanoma | interventions — reolysin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (viral therapy) (Experimental): Patients receive wild-type reovirus (Reolysin®) IV administered at a dose of 3 x 10^10 TCID50/day in 250 mL 0.9% sodium chloride infused intravenously over 60 minutes daily on days 1-5 of each 28-day cycle. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: wild-type reovirus

INTERVENTIONS:
Biological: wild-type reovirus — Given IV: Administered at a dose of 3 x 10^10 TCID50/day in 250 mL 0.9% sodium chloride infused intravenously over 60 minutes daily on days 1-5 of each 28-day cycle.
  Other Names: REOLYSIN

SUMMARY:
This phase II trial is studying the side effects and how well viral therapy works in treating patients with metastatic melanoma. Viral therapy may be able to kill tumor cells without damaging normal cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Assess the antitumor effect of wild-type reovirus (Reolysin®), in terms of tumor response rate and clinical benefit rate (i.e., partial response and complete response), in patients with metastatic melanoma.

II. Assess the toxicity profile of Reolysin® in these patients.

SECONDARY OBJECTIVES:

I. Assess the progression-free survival and overall survival of these patients. II. Assess viral replication in metastatic melanoma deposits after intravenous administration of Reolysin®.

III. Assess the impact of pre-existing anti-reoviral immunity (as represented by p38 expression in pretreatment tumor specimens) on the efficacy and toxicity of Reolysin®.

IV. To measure the effect of Reolysin® on the immune system, in terms of dendritic cell activation, T-cell activation, presence of Treg cells in tumor specimens, and the frequency of T cells, B cells, NK cells, and peptide specific cytotoxic T lymphocytes reactive against melanoma differentiation antigen peptides (gp100, MART-1, and tyrosinase).

V. To assess the induction of melanoma specific immune response, in terms of the presence of melanoma differentiation antigens (gp100, MART-1, and tyrosinase) in tumor specimens.

OUTLINE: This is a multicenter study.

Patients receive wild-type reovirus (Reolysin®) IV over 60 minutes on days 1-5. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.

Some patients undergo tumor tissue samples collection at baseline and at 1 week after initiation of treatment for correlative laboratory studies. Tissue samples are analyzed for p38/MAPK activation status by IHC; reoviral replication in metastatic deposits by electron microscopy; and immunologic parameters by IHC. Blood samples are collected at baseline and periodically during the study. Blood samples are analyzed for immunologic parameters by tetramer and ELISPOT technology and for neutralizing antibodies against reovirus.

After completion of study treatment, patients are followed every 6 months for 2 years and then annually for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed malignant melanoma

  * All melanomas, regardless of origin, are allowed
  * Metastatic disease
* Measurable disease, defined as ≥ 1 lesion that can be accurately measured in ≥ 1 dimension (longest diameter to be recorded) as ≥ 20mm by conventional techniques or as ≥ 10 mm by spiral CT scan
* Must have ≥ 1 metastatic lesion that can be safely biopsied
* Must have received ≥ 1 prior treatment for metastatic disease
* Not a candidate for curative surgery for metastatic disease
* No known brain metastases
* Eastern Cooperative Oncology Group performance status 0-2
* Life expectancy > 12 weeks
* Total White Blood Cell (WBC) ≥ 3,000/mcL
* Absolute neutrophil count ≥ 1,500/mcL
* Platelet count ≥ 100,000/mcL
* Hemoglobin ≥ 9 g/dL
* Total bilirubin ≤ 1.5 times upper limit of normal (ULN)
* Aspartate Aminotransferase (AST) ≤ 2.5 times ULN
* Creatinine ≤ 1.5 times ULN
* Troponin-T normal
* Left ventricular ejection fraction (LVEF) ≥ 50% by ECHO or MUGA
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Agrees to provide blood and tissue samples for the mandatory translational research component of the study
* Must be able to avoid direct contact with pregnant or nursing women, infants, and immuno compromised individuals during study and for ≥ 3 weeks following the last dose of study agent
* No concurrent uncontrolled illness including, but not limited to, any of the following:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris, cardiac arrhythmia, or myocardial infarction within the past year
  * Psychiatric illness/social situation that would preclude study compliance
* No known HIV positivity

  * Patients with a clinical history suggestive of an immuno compromised status are required to undergo HIV testing
* More than 4 weeks since prior chemotherapy (6 weeks for mitomycin C or nitrosoureas) and recovered
* More than 2 weeks since prior radiotherapy, immunotherapy, or treatment with small molecule cell cycle inhibitors
* No other concurrent investigational agents
* No other concurrent anticancer therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2008-04; Primary Completion 2011-12 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Evanthia Galanis, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Twenty three participants were enrolled onto this study between August 2008 and January 2010.
Pre-assignment Details: One participant died prior to receiving any treatment and is not included in this study summary. One participant was found to be ineligible and was not used in the analysis of any endpoint, but was used for reporting toxicity. Therefore, 21 participants were used for the primary analysis and 22 participants are used to report toxicity.
Groups:
- Treatment (Viral Therapy): Patients receive wild-type reovirus (Reolysin®) IV over 60 minutes on days 1-5. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Treatment (Viral Therapy)
Started | 23
Completed | 21
Not Completed | 2
Not completed — Death | 1
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Viral Therapy)
Number analyzed (Participants) | 21
Age, Continuous [Median (Full Range); unit: years] | 65 [22 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 9
Region of Enrollment [Number; unit: participants]
  United States | 21

OUTCOME MEASURES:

1. Primary Outcome: Tumor Response
Description: A tumor response is defined to be a Complete Response (CR) or Partial Response (PR) as defined by the Response Evaluation Criteria in Solid Tumors (RECIST) noted as the objective status on 2 consecutive evaluations at least 4 weeks apart.
  Complete Response (CR): Disappearance of all target lesions. Partial Response (PR): At least a 30% decrease in the sum of the largest dimension (LD) of target lesions taking as reference the baseline sum LD.
Time Frame: Every 4 weeks after 4 courses of treatment, assessed up to 5 years
Measure: Number; unit: participants
Arm/Group | Treatment (Viral Therapy)
Number analyzed (Participants) | 21
participants
  Complete Response (CR) | 0
  Partial Response (PR) | 0

2. Secondary Outcome: Overall Survival
Description: Survival time is defined as the time from registration to death due to any cause. The distribution of survival time will be estimated using the method of Kaplan-Meier.
Time Frame: Time from registration to death due to any cause, assessed up to 5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Viral Therapy)
Number analyzed (Participants) | 21
months | 5.42 [0.49 to 15.8]

3. Secondary Outcome: Time to Disease Progression
Description: Time to disease progression is defined as the time from registration to documentation of disease progression. If a patient dies without documentation of disease progression, the patient will be considered to have had tumor progression at the time of their death unless there is sufficient documented evidence to conclude no progression occurred prior to death.
Time Frame: Time from registration to documentation of disease progression, assessed up to 5 years
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Treatment (Viral Therapy)
Number analyzed (Participants) | 21
days | 45 [13 to 96]

ADVERSE EVENTS:
Arm/Group | Treatment (Viral Therapy)
Serious Adverse Events (participants affected / at risk) | 11/22
Other Adverse Events (participants affected / at risk) | 22/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Viral Therapy) (N=22)
Hemoglobin decreased (Blood and lymphatic system disorders) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Left ventricular failure (Cardiac disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Disease progression (General disorders) | 1 (1)
Fatigue (General disorders) | 2 (2)
Fever (General disorders) | 1 (1)
Alkaline phosphatase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Laboratory test abnormal (Investigations) | 1 (1)
Leukocyte count decreased (Investigations) | 2 (2)
Lymphocyte count decreased (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 2 (3)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Blood uric acid increased (Metabolism and nutrition disorders) | 1 (1)
Serum albumin decreased (Metabolism and nutrition disorders) | 4 (5)
Serum calcium decreased (Metabolism and nutrition disorders) | 2 (2)
Serum calcium increased (Metabolism and nutrition disorders) | 1 (1)
Serum phosphate decreased (Metabolism and nutrition disorders) | 2 (2)
Serum sodium decreased (Metabolism and nutrition disorders) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 1 (1)
Ischemia cerebrovascular (Nervous system disorders) | 1 (1)
Confusion (Psychiatric disorders) | 2 (2)
Insomnia (Psychiatric disorders) | 1 (1)
Ureteric obstruction (Renal and urinary disorders) | 1 (1)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hemorrhage (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Viral Therapy) (N=22)
Hemoglobin decreased (Blood and lymphatic system disorders) | 16 (27)
Diarrhea (Gastrointestinal disorders) | 4 (6)
Nausea (Gastrointestinal disorders) | 12 (16)
Vomiting (Gastrointestinal disorders) | 6 (6)
Chills (General disorders) | 11 (16)
Fatigue (General disorders) | 19 (29)
Fever (General disorders) | 11 (18)
Leukocyte count decreased (Investigations) | 6 (9)
Lymphocyte count decreased (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 2 (2)
Platelet count decreased (Investigations) | 9 (11)
Anorexia (Metabolism and nutrition disorders) | 12 (17)
Serum sodium decreased (Metabolism and nutrition disorders) | 1 (1)
Joint pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 12 (14)
Headache (Nervous system disorders) | 3 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (11)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 (7)
Rash desquamating (Skin and subcutaneous tissue disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less